CLINICAL TRIAL: NCT06536933
Title: Study of Metabolic Dysfunction-Associated Steatotic Liver Disease Among Sohag University Employees
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Eldin Hamdy Hamed, Resident-Internal Medicine department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-07-19MS
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Abdominal Ultrasound — Diagnostic non invasive Abdomibal Ultrasound will be done to quantify hepatic steatosis

SUMMARY:
* Metabolic dysfunction-associated steatotic liver disease (MASLD) is the latest term for steatotic liver disease associated with metabolic syndrome. MASLD is a common cause of chronic liver disease and is the leading cause of liver-related morbidity and mortality.
* The high prevalence of this disease has been fueled by the rapid rise in levels of sedentary behavior, low levels of physical activity, excess calorie intake relative to expenditure in nutritionally imbalanced and unhealthy diets. In parallel, the prevalence of poor metabolic health in adults from many countries is high, even in normal weight individuals.
* MASLD has been estimated to affect 30% of the adult population worldwide, with its prevalence increasing from 22% to 37% from 1991 to 2019 . The increasing prevalence of MASLD parallels the increasing prevalence of obesity and obesity-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* 100 Employees in Sohag University will be included in the study.

Exclusion Criteria:

Employees with drug induced liver disease. Employees with chronic liver disease. Employees with decompensated liver cirrhosis. Employees with excessive alcohol consumption.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 100 Employees in Sohag University will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
waist circumference | 4 months
  by using a flexible non-stretchable measuring tape by identifying measurement point midway between the lower margin of last palpable rib and the top of iliac crest.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan WK, Chuah KH, Rajaram RB, Lim LL, Ratnasingam J, Vethakkan SR. Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A State-of-the-Art Review. J Obes Metab Syndr. 2023 Sep 30;32(3):197-213. doi: 10.7570/jomes23052. Epub 2023 Sep 13. PMID 37700494
- [Background] Inoue Y, Qin B, Poti J, Sokol R, Gordon-Larsen P. Epidemiology of Obesity in Adults: Latest Trends. Curr Obes Rep. 2018 Dec;7(4):276-288. doi: 10.1007/s13679-018-0317-8. PMID 30155850
- [Background] Stefan N, Schick F, Haring HU. Causes, Characteristics, and Consequences of Metabolically Unhealthy Normal Weight in Humans. Cell Metab. 2017 Aug 1;26(2):292-300. doi: 10.1016/j.cmet.2017.07.008. PMID 28768170
- [Background] Chan WK, Treeprasertsuk S, Imajo K, Nakajima A, Seki Y, Kasama K, Kakizaki S, Fan JG, Song MJ, Yoon SK, Dan YY, Lesmana L, Ho KY, Goh KL, Wong VW. Clinical features and treatment of nonalcoholic fatty liver disease across the Asia Pacific region-the GO ASIA initiative. Aliment Pharmacol Ther. 2018 Mar;47(6):816-825. doi: 10.1111/apt.14506. Epub 2018 Jan 14. PMID 29333610